CLINICAL TRIAL: NCT01852968
Title: Hippocampal Metabolism and Function in Patients With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1301M26901
Record Dates: First submitted 2013-04-12; First posted 2013-05-14 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Hypoglycemia; Diabetes Mellitus
Keywords: hypoglycemia; hypoglycemia unawareness; type 1 diabetes, hippocampus; glucose transport; cognitive dysfunction
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus; Diabetes Mellitus, Type 1; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood smaple will be drawn measurement of blood glucose, HgbA1C, insulin and hormone levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with type 1 diabetes: Hippocampal neurochemistry and metabolism will examined in Patients with type 1 diabetes using magnetic resonance spectroscopy.
  Patients with type 1 diabetes will also undergo neurocognitive testing to assess hippocampal function
- healthy controls: Hippocampal neurochemistry and metabolism will be examined in healthy controls using magnetic resonance spectroscopy.
  Healthy controls will also undergo neurocognitive testing to assess hippocampal function

SUMMARY:
The hippocampus is an area of brain which plays an essential role in learning and memory processing and is thought to be particularly vulnerable to effects of hypoglycemia (low blood glucose). The goal of this project is to examine hippocampal neurochemistry and metabolism and identify how diabetes and recurrent hypoglycemia alter the hippocampus.

DETAILED DESCRIPTION:
In this study we will examine hippocampal neurochemical profile and glucose transport kinetics using magnetic resonance spectroscopy (MRS) in patients with type 1 diabetes and hypoglycemia unawareness and matched healthy controls. We will also examine hippocampal function in these subject groups during euglycemia and hypoglycemia and correlate these findings to changes in the neurochemical profile and glucose transport kinetics.

Study protocol

MRS experiments On the morning of the MRS experiments, subjects will present to the Center for Magnetic Resonance Research (CMRR) at 7 AM in the fasting state to participate in a protocol with which our group has significant experience. After arrival, they will be prepared for the clamp study by the placement of one intravenous catheter into one vein in antecubital fossa for the later infusion of glucose, insulin, and potassium. A second intravenous catheter will be placed retrograde into a vein in the distal leg for later blood sampling. An intravenous infusion of insulin will then be started and adjusted as necessary to bring blood glucose to 95 mg/dl. Blood will be collected every 10 minutes for measurement of glucose on a nearby Analox machine to guide adjustments in the insulin infusion rate. The experiment will begin when the subject is at 95 mg/dl. At time 0, the intravenous insulin infusion will be fixed at 1 mU/kg/min, samples for blood glucose will be collected every 5 minutes and an intravenous infusion of glucose (20% dextrose) will be administered as necessary to maintain blood glucose at 95 mg/dl. At +5 minutes, subjects will be placed into the magnet. Blood glucose will be maintained at 95 mg/dl during the next 25 minutes as the hippocampal volume-of-interest (VOI) is selected and baseline MRS data are acquired. At + 30 min, subjects will be given an intravenous bolus injection of glucose over 1-2 minutes using the formula of administering 2 mg glucose/kg body weight for each 1 mg/dl increase desired that our group have used with success previously. Immediately after the bolus injection, a continuous infusion of 20% dextrose will be started and the rate of administration will be adjusted to maintain the desired glucose target of 200 mg/dl, 300 mg/dl, or 400 mg/dl. MRS data will be collected continuously starting 10 minutes before the bolus injection (baseline) until the end of the study ~60 minutes after the bolus, which is sufficient to reach steady-state glucose concentrations in the brain and maintain them for at least 20 minutes. At the completion of the study, the infusions will be discontinued; the subject will resume their usual insulin regimen, and be fed a meal. The subjects with diabetes will be prepared for this protocol by instructing them to manage their diabetes in such a way as to minimize the amount of subcutaneous insulin present at the time of the study without creating hyperglycemia on the day before the study (i.e. pump patients will stop their pump on arrival, glargine treated patients will take last glargine dose 24 hours before study start). At the conclusion of the study, subjects will be allowed to resume their usual insulin regimen.

Neurocognitive testing On the morning of the Neurocognitive testing, subjects will present to the Clinical and Translational Science Institute at 7 AM in the fasting state. Subjects with diabetes will have their blood glucose checked to ensure that blood glucose is between 90-200 mg/dl. If the blood glucose is not in target range, treatment will be given to correct glucose or the study will be rescheduled. Subjects will undergo neurocognitive testing with the California Verbal Learning Test - Second Edition (CVLT-II) and subtests from the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): Story Memory (immediate and delayed), Digit Span, and Coding. After completion of neurocognitive testing, an intravenous catheter will be placed antegrade in each forearm for subsequent infusions and for blood sampling. Insulin will be infused at a rate of 2.0 mU/kg/min along with potassium phosphate (4 mEq/hour) and blood glucose will reduced to and then maintained at 55 mg/dl by the variable infusion of 20% dextrose. Samples for blood glucose will be collected every 5 minutes for measurement of glucose. Once the blood glucose target of 55 is achieved subject will undergo neurocognitive testing again. At the completion of the neurocognitive testing subjects will be fed and euglycemia will be restored.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of type 1 diabetes, hemoglobin A1C <9%. Alternatively, subject should be a healthy control.

Exclusion Criteria:

Exclusion criteria for both groups of subjects include history of stroke, seizures, neurosurgical procedures, or arrhythmias, and use of drugs that can alter glucose metabolism (other than insulin for the patients with diabetes). Subjects must also meet requirements for a study in the magnet, which includes weight less than 300 lbs. and the absence of metallic substances in their body.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University of Minnesota Endocrine Clinic, univeristy of Minnesota community and a registry of volunteers maintained by the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-05; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
alterations in hippocampal glucose transport kinetics | data will be acquired at the time of experiment.
  Hippocampal glucose transport kinetics will be examined using magnetic resonance spectroscopy

SECONDARY OUTCOMES:
hippocampal function | data will be collected on day of experiment
  Subjects will undergo neurocognitive testing with the California Verbal Learning Test - Second Edition (CVLT-II)and subtests from the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS: Story Memory (immediate and delayed), Digit Span, and Coding.
alterations in hippocampal neurochemistry | data will be acquired at the time of experiment
  Hippocampal neurochemical profile will be examined using magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Amir Moheet, MD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Science Institute and Center for Magnetic Resonance Research, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Bednarik P, Henry PG, Khowaja A, Rubin N, Kumar A, Deelchand D, Eberly LE, Seaquist E, Oz G, Moheet A. Hippocampal Neurochemical Profile and Glucose Transport Kinetics in Patients With Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Feb 1;105(2):479-91. doi: 10.1210/clinem/dgz062. PMID 31637440